CLINICAL TRIAL: NCT03175276
Title: Predict IQCODE Delirium in Geriatric Patients
Brief Title: Informant Questionaire on Cognitive Decline in the Elderly (IQCODE) and Delirium in Geriatric Patients
Acronym: Delirium
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Other Study IDs: Cognitive decline and delirium
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2017-03

CONDITIONS: Delirium in Old Age; Cognitive Decline
Keywords: Delirium; Cognitive decline; IQCODE
MeSH Terms: conditions — Cognitive Dysfunction; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the usefulness of the Informant Questionaire on Cognitive Decline in the Elderly (IQCODE) to predict delirium in elderly patients admitted to Emergency Department (ED) with geriatric assessment and transferred to Geriatric ward.

DETAILED DESCRIPTION:
Design: The project will be conducted as a prospective study.

Methods:

Exposure: The short IQCODE is a 16-item questionnaire that ask relatives about changes in the elderly patients cognitive performance over the previous 10 years. The score range from one to five, with a high score reflecting bad evolution through the years.

Settings: Patients (aged ≥75 years) admitted to ED (medical and surgery) and transferred to a geriatric ward at Aarhus University Hospital, who meet the inclusion criteria will be asked if the staff is allowed to contact their relatives. By oral consent, the relatives are interviewed by telephone or at the hospital. The IQCODE are filled in during the interview.

In the geriatric ward the assessment of delirium by a positive Confusion Assesment Method (CAM) is done twice a day and is part of the regular procedure in the Geriatric Department at Aarhus University Hospital.

Sample size: The power calculation is based on a pilot study of IQCODE. The study that included 32 75-year-olds from geriatric ward at Aarhus University hospital, showed an no incidence of delirium of when the IQCODE-score was ≤3,125. On the contrary the incidence of delirium was 15% when the IQCODE-score was >3,125. With a power of 90% and a significance level of 5%, 76 patients should be included in each group to predict delirium.

Time frame: Of the 80 admitted to the geriatric wards, only 20% in the pilot study had an IQCODE-score ≤3,125. With an expected response rate of 70%, the data collection period is expected to last five months.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the emergency medical and surgery ward and transferred to a geriatric ward at Aarhus University Hospital in the period from the 20th of March to September 2017.

Exclusion Criteria:

* Patients transferred to the geriatric ward in the evening and night as well as weekends and holidays, when there is no Geriatric staff present.
* Patients who upon admission are dying assessed by a geriatrician
* Patients with stroke where aphasia is present
* Patients with severe dementia without language
* Patients who are inability to understand or speak Danish

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients (aged ≥75 years), acutely admitted to ED and transferred to a geriatric ward at Aarhus University Hospital in the period from March to September 2017 for diseases that need either medical or surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Delirium | Repeated measurements twice a day at 7-11 AM and 5-10 PM until discharge
  Delirium diagnosed using the Confusion Assessment Method (CAM) - Danish version. Incidence of delirium is measured by the first positive CAM score.

CONTACTS AND LOCATIONS:
Overall Officials: Else Marie Damsgaard, Professor, Study Chair — Department of Geriatrics , Aarhus University Hospital Palle Juul-Jensens Boulevard 99, Building J, J513, DK-8200 Aarhus N
Locations (1):
- Aarhus University hospital, Aarhus, Central Danmark Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Priner M, Jourdain M, Bouche G, Merlet-Chicoine I, Chaumier JA, Paccalin M. Usefulness of the short IQCODE for predicting postoperative delirium in elderly patients undergoing hip and knee replacement surgery. Gerontology. 2008;54(2):116-9. doi: 10.1159/000117574. Epub 2008 Feb 18. PMID 18285677
- [Background] Siddiqi N, Harrison JK, Clegg A, Teale EA, Young J, Taylor J, Simpkins SA. Interventions for preventing delirium in hospitalised non-ICU patients. Cochrane Database Syst Rev. 2016 Mar 11;3(3):CD005563. doi: 10.1002/14651858.CD005563.pub3. PMID 26967259